CLINICAL TRIAL: NCT03106935
Title: Effect of Levothyroxine Treatment on Pregnancy Outcome in RPL Women With Subclinical Hypothyroidism
Brief Title: Recurrent Pregnancy Loss and Thyroid Disease
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Second Affiliated Hospital of Soochow University (Other)
Responsible Party: Principal Investigator, ZHANG Hong, Ph.D,M.D, Second Affiliated Hospital of Soochow University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: The Second Affiliated Hospital
Record Dates: First submitted 2017-02-27; First posted 2017-04-11 (Actual); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Recurrent Pregnancy Loss
Keywords: recurrent pregnancy loss; Clinical hypothyroidism; Subclinical hypothyroidism; thyroid stimulating hormone; thyroid peroxidase antibody; Levothyroxine
MeSH Terms: interventions — Thyroxine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (2):
- Obstet Gynecol,SecondSoochowU (Active Comparator): Levothyroxine is an orodispersible tablet.For the LT4 treatment group, 50μg LT4 (Merck Serono, Geneva,Switzerland) was administered every morning from the first day of diagnosed as subclinical hypothyroidism and continued up to the day of serum β-HCG measurement.If pregnancy was confirmed, levothyroxine dose need to increase 25-30% and adjusted according to the pregnancy specific reference range ( T1 0.1-2.5mIU/L,T2 0.2-3.0mIU/L, T3 0.3-3.0mIU/L) .
  Interventions: Drug: Levothyroxine
- reproductive center,SecondSoochowU (No Intervention): For the control group ,women with subclinical hypothyroidism are not given any drugs .

INTERVENTIONS:
Drug: Levothyroxine — Levothyroxine is an orodispersible tablet.For the LT4 treatment group, 50μg LT4 (Merck Serono, Geneva,Switzerland) was administered every morning from the first day of diagnosed as subclinical hypothyroidism and continued up to the day of serum β-HCG measurement.If pregnancy was confirmed, levothyroxine dose need to increase 25-30% and adjusted according to the pregnancy specific reference range ( T1 0.1-2.5mIU/L,T2 0.2-3.0mIU/L, T3 0.3-3.0mIU/L) .
  Other Names: LT4
  Arms: Obstet Gynecol,SecondSoochowU

SUMMARY:
The present study is divided into two groups ,one is the patients with subclinical hypothyroidism who has TPO antibody positive women with TSH concentrations > 2.5 mU/L and below the upper limit of the pregnancy specific reference range ,another is TPO antibody negative with TSH concentrations greater than the pregnancy specific reference range and below 10.0 mU/L.The two groups are randomized into either the LT4 treatment group or control group by the use of a computer-generated list.

The aim of our study is to determine whether the use of levothyroxine is beneficial in patients with subclinical hypothyroidism in two groups。

DETAILED DESCRIPTION:
Many studies have stratified the risk imparted by hypothyroidism according to TPOAb status, and consistently show that this risk is higher in TPOAb positive women. Some data also suggest that the adverse impact associated with maternal TSH levels is apparent at lower TSH elevations in women known to be TPOAb positive compared to women who are TPOAb negative. Furthermore, studies suggest a reduction in pregnancy loss when TPOAb positive women are treated with levothyroxine, even when biochemically euthyroid. Intervention trials have not been performed in TPOAb negative women. A etiology analysis process,from June 2010 to June 2015 in The Second Affiliated Hospital of Soochow University, were showed that 22.2% of total 917 cases who had RPL history present as abnormal serum TSH level or positive TPOAb, while 36.6% of 523 cases who repregnancy present as abnormal.This present study is divided into two groups ,one is the patients with subclinical hypothyroidism who hasTPO antibody positive women with TSH concentrations > 2.5 mU/L and below the upper limit of the pregnancy specific reference range ,another is TPO antibody negative with TSH concentrations greater than the pregnancy specific reference range and below 10.0 mU/L.The two groups are randomized into either the LT4 treatment group or control group by the use of a computer-generated list.For the LT4 treatment group, 50μg LT4 (Merck Serono, Geneva,Switzerland) was administered every morning from the first day of diagnosed as subclinical hypothyroidism and continued up to the day of serum β-HCG measurement.If pregnancy was confirmed, levothyroxine dose need to increase 25-30% and be adjusted according to the pregnancy specific reference range ( T1 0.1-2.5mIU/L,T2 0.2-3.0mIU/L, T3 0.3-3.0mIU/L).For the control group ,women with subclinical hypothyroidism are not given any drugs . The aim of our study is to determine whether the use of levothyroxine is beneficial in patients with subclinical hypothyroidism who has TPO antibody positive women with TSH concentrations > 2.5 mU/L and below the upper limit of the pregnancy specific reference range or TPO antibody negative with TSH concentrations greater than the pregnancy specific reference range and below 10.0 mU/L.

ELIGIBILITY:
Inclusion Criteria:

1. having a diagnosis of RPL (two or more consecutive or non-consecutive first-trimester losses)
2. be.ing aged 18-39 years at randomisation
3. trying to conceive naturally
4. willing and able to give informed consent

Exclusion Criteria:

1. they were unable to conceive naturally (as confirmed by urinary pregnancy tests) within 1 year of recruitment or before the end of the randomisation period in the trial, whichever came earlier
2. they had antiphospholipid syndrome [lupus anticoagulant and/or anticardiolipin antibodies (immunoglobulin G or immunoglobulin M)]; other recognised thrombophilic conditions (testing according to usual clinic practice) l they had uterine cavity abnormalities (as assessed by ultrasound, hysterosonography, hysterosalpingogram or hysteroscopy)
3. they had abnormal parental karyotype
4. they had other identifiable causes of RPL (tests initiated only if clinically indicated) such as diabetes or systemic lupus erythematosus
5. they had any contraindications to Levothyroxine use

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2015-07; Primary Completion 2017-12 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Gestational week at delivery | 28 weeks
  The research doctor site telephoned every participant 2 weeks after the expected date of delivery to obtain pregnancy outcome data.
Newborn birth weight | at birth
  The research doctor site telephoned every participant 2 weeks after the expected date of delivery to obtain newborn birth weight.
APGAR Score at birth | at birth
  The APGAR (Appearance, Pulse, Grimace, Activity, Respiration) scale is determined by evaluating the newborn baby on five simple criteria on a scale from zero to two, then summing up the five values thus obtained. The resulting APGAR score ranges from zero to 10.

SECONDARY OUTCOMES:
Number of clinical pregnancy at 6-8 weeks (defined as the presence of a gestational sac, with or without a yolk sac or fetal pole) | 8 weeks
  The research doctor site telephoned every participant at between 6 and 7 weeks of gestation, to ensure there were arrangements for an ultrasound appointment with her usual carers, before 8 weeks of gestation. If an appointment had not been booked, the research doctor assisted with booking. The research doctor telephoned each participant again between 3 and 5 days after the scheduled date of the ultrasound appointment, to obtain details of the observations of a gestational sac.
Number of ongoing pregnancy at 12 weeks (defined as the presence of a fetal heartbeat) | 12weeks
  The research doctor site telephoned each participant between 10 and 12 weeks of gestation, to ensure there were arrangements for an ultrasound appointment with her usual carers, at between 12 and 14 weeks of gestation. As previously, the research doctor assisted with booking an appointment if necessary, and telephoned the participant afterwards to obtain details of variables such as fetal heartbeat. The research doctor also recorded the expected date of delivery at this stage.
Number of miscarriage (defined as loss of pregnancy before 28 weeks of gestation). | 28 weeks
  The research doctor site telephoned each participant before28 weeks of gestation, to obtain their pregnancy outcomes such as miscarriage.

CONTACTS AND LOCATIONS:
Overall Officials: ZHANG Hong, Ph.D,M.D, Principal Investigator — a staff of The Second Affiliated Hospital of Soochow University
Locations (1):
- Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zhu LY, Chen X, Xu ZZ, Xu L, Mao T, Zhang H. Changes and clinical significance of peripheral blood helper T lymphocyte and natural killer (NK) cells in unexplained recurrent spontaneous abortion (URSA) patients after abortion and successful pregnancy. Clin Exp Obstet Gynecol. 2015;42(1):62-6. PMID 25864284
- [Background] Wu S, Zhang H, Tian J, Liu L, Dong Y, Mao T. Expression of kisspeptin/GPR54 and PIBF/PR in the first trimester trophoblast and decidua of women with recurrent spontaneous abortion. Pathol Res Pract. 2014 Jan;210(1):47-54. doi: 10.1016/j.prp.2013.09.017. Epub 2013 Oct 26. PMID 24225150
- [Background] Zhang H, Long Q, Ling L, Gao A, Li H, Lin Q. Elevated expression of KiSS-1 in placenta of preeclampsia and its effect on trophoblast. Reprod Biol. 2011 Jul;11(2):99-115. doi: 10.1016/s1642-431x(12)60048-5. PMID 21804632
- [Background] Mao C, Zhang H, Xiao D, Zhu L, Ding Y, Zhang Y, Wu L, Xu Z, Zhang L. Perinatal nicotine exposure alters AT 1 and AT 2 receptor expression pattern in the brain of fetal and offspring rats. Brain Res. 2008 Dec 3;1243:47-52. doi: 10.1016/j.brainres.2008.09.060. Epub 2008 Oct 2. PMID 18926802